CLINICAL TRIAL: NCT04643730
Title: Randomised Controlled Study: The Effects on Pain of Foot Reflexology and Acupressure During Heel Lancing In Newborns
Brief Title: The Effects on Pain of Acupressure and Foot Reflexology Before Heel Lancing in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayşe Özge DENİZ, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Ayşe Özge DENİZ
Record Dates: First submitted 2020-10-10; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Interventions Pain
Keywords: Newborn,; pain,; heel lance,; foot reflexology,; acupressure,; nurse
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reflexology Group (Experimental): Foot Reflexology was applied to the babies before heel lancing
  Interventions: Other: Foot Reflexology Methods
- Acupressure Group (Experimental): Acupressure was applied to the babies before heel lancing
  Interventions: Other: Acupressure methods
- Control Group (Active Comparator): No pre-application was made to the babies in the control group as a routine procedure
  Interventions: Other: Control Grup

INTERVENTIONS:
Other: Acupressure methods — Acupressure on the KI3 and St36 points applied to the babies in the acupressure group for a total of 7 minutes before the heel prick
  Arms: Acupressure Group
Other: Foot Reflexology Methods — Foot reflexology was applied to the babies in the foot reflexology group for a total of 7 minutes before the heel prick
  Arms: Reflexology Group
Other: Control Grup — No pre-application was made to the babies in the control group as a routine procedure.
  Arms: Control Group

SUMMARY:
This study aimed to determine the effects of foot reflexology and acupressure on the KI3 and St36 points on pain during interventions when these procedures were administered before heel lancing in term newborns.

ELIGIBILITY:
Inclusion Criteria:

1. Being born by cesarean section,
2. Being a term newborn,
3. Being completed the 24th hour of the postnatal period,
4. Staying with birth mother,
5. Being fed in the last half hour before the procedure,
6. Having a heel prick performed by the same nurse,
7. Giving blood on the first try (because pain level may change on the second try),
8. Having a mother who gave written informed consent

Exclusion Criteria:

1. Having no health problem,
2. Being underwent more than 2 invasive interventions,
3. Receiving an analgesic/sedative drug in the 8 hours before the application.

Min Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Pain levels of the newborns | Before the pain procedure, during the pain procedure (the pain levels of the infants when the needle pricked the heel were evaluated using the N-PASS) and After the pain procedure. (Having completed the 24th hour of the postnatal period)
  The N-PASS was developed by Hummel et al. in 2003 to be used in all full-term and preterm neonates. The scale was revised by Hummel on October 2, 2009 and adapted to Turkish by Açıkgöz et al. in 2011 The Cronbach's alpha internal consistency coefficient of the scale was found to be 0.779 for preintervention and 0.917 for postintervention (Açıkgöz et al., 2017). The N-PASS consists of five sub-dimensions: crying and irritability, behavior-state, facial expression, extremities tone, and vital signs. The sub-dimension of vital signs was evaluated according to infants' heart rates and oxygen saturation values. The total pain score that can be obtained from the scale ranges between 0 and +10. A higher score indicates that the severity of pain is high. The goal of pain therapy is to keep the score at or below 3 (Hummel et al., 2008; Hummel et al., 2010).

SECONDARY OUTCOMES:
Changes in oxygen saturation | 2 Minutes
  Recorded the changes in oxygen saturation (SpO2) of newborns (Having completed the 24th hour of the postnatal period) before (A pulse oximeter was attached to the infants two minutes before the procedure), during and after pain procedure
Changes in heart rates | 2 Minutes
  Recorded the changes in Heart rate of newborns (Having completed the 24th hour of the postnatal period) before (A pulse oximeter was attached to the infants two minutes before the procedure), during and after pain procedure
Percentage of crying during heel prick in healthy term neonates | During heel prick and immediately after intervention
  Percentage of crying in 3 groups were applied during heel prick and immediately after intervention. Results are shown as mean.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Public Hospital, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830
- [Background] Hummel P, Lawlor-Klean P, Weiss MG. Validity and reliability of the N-PASS assessment tool with acute pain. J Perinatol. 2010 Jul;30(7):474-8. doi: 10.1038/jp.2009.185. Epub 2009 Nov 19. PMID 19924132
- [Background] Açıkgöz, A., Çiğdem, Z., Yıldız, S., Demirüstü, C., Yarar, M., & Aksit, A. (2017). A Turkish Adaptation of the Neonatal Pain/Agitation, Sedation Scale (N-PASS) and its Validity and Reliability, Indian Journal of Fundamental and Applied Life Sciences, 7(2): 5-11
- [Derived] Deniz AO, Acikgoz A. A Randomized Controlled Trial: The Effect of Acupressure and Foot Reflexology on Pain During Heel-Lancing in Neonates. Clin Nurs Res. 2023 Feb;32(2):306-312. doi: 10.1177/10547738211061815. Epub 2021 Dec 26. PMID 34955035